CLINICAL TRIAL: NCT01891305
Title: A Phase 2a, Randomized, Double-Blind, Placebo-Controlled, Dose Ranging Study to Evaluate the Efficacy and Safety of VT-1161 Oral Tablets in the Treatment of Patients With Moderate to Severe Interdigital Tinea Pedis
Brief Title: A Study to Evaluate the Efficacy and Safety of Oral VT-1161 in Patients With Moderate - Severe Interdigital Tinea Pedis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Viamet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VMT-VT-1161-CL-003
Record Dates: First submitted 2013-06-17; First posted 2013-07-03 (Estimated); Results first posted 2018-07-06 (Actual); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Tinea Pedis
MeSH Terms: conditions — Tinea Pedis | interventions — VT-1161

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- VT-1161 200/50mg (Experimental)
  Interventions: Drug: VT-1161
- VT-1161 600/150mg (Experimental)
  Interventions: Drug: VT-1161
- VT-1161 1200/300mg (Experimental)
  Interventions: Drug: VT-1161
- Matching placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: VT-1161
  Arms: VT-1161 1200/300mg; VT-1161 200/50mg; VT-1161 600/150mg
Drug: placebo
  Arms: Matching placebo

SUMMARY:
The purpose of this study is to determine if the novel oral agent VT-1161 is safe and effective in treating patients with moderate - severe tinea pedis (also referred to as athletes foot). VT-1161 has been designed to inhibit CYP51, an enzyme essential for fungal growth. Inhibition of CYP51 results in the accumulation of chemicals know to be toxic to the fungus. CYP51 is the molecular target of the class of drugs referred to as 'azole antifungals'. All currently approved azole drugs have poor selectivity for CYP51 and this results in many of the side effects associated with the azole antifungals. The safety profile of the class similarly limits use in chronic treatment of non-life-threatening fungal infections. A safer antifungal drug would improve treatment options for infections seen in otherwise healthy individuals where significant side-effect risks are unacceptable.

ELIGIBILITY:
Key Inclusion Criteria:

* Healthy male and non-pregnant female patients ≥18 years and <65 years
* Clinical diagnosis of tinea pedis
* Positive baseline KOH
* Clinical signs and symptoms score of the target lesion is at least 6, including a minimum score of at least 2 for erythema AND a minimum score of 2 for either scaling or pruritus (on a scale of 0-3, where 2 indicates moderate severity)
* Patients must be able to swallow capsules intact
* Use acceptable birth control methods

Key Exclusion Criteria:

* Major organ system disease or clinical infection
* Poorly controlled diabetes mellitus
* Pregnant or lactating
* Confluent, diffuse moccasin-type tinea pedis
* Presence of onychomycosis involving a) more than 5 toe nails, b) any fingernail
* Recent use of topical corticosteroids, topical antibiotics, or topical antifungal therapy to the foot
* Recent use of systemic corticosteroids or antifungal therapy
* Known(HIV)infection
* Known significant hepatic, or hematologic impairment .Requirement for treatment with concomitant antimicrobial or systemic antifungal therapy for any reason.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-08; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Univ Alabama at Birmingham, Birmingham, Alabama
  - Florida Academic Dermatology Center, Miami, Florida
  - FXM Research, Miramar, Florida
  - Wake Research Associates, Raleigh, North Carolina
  - Oregon Dermatology & Research Center, Portland, Oregon
  - J&S Studies, Inc., College Station, Texas
  - Pariser Dermatology Specialists, Norfolk, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- VT-1161 200/50mg: VT-1161 200mg once daily for 4 days, then VT-1161 50mg once daily for 10 days
- VT-1161 600/150mg: VT-1161 600mg once daily for 4 days, then VT-1161 150mg once daily for 10 days
- VT-1161 1200/300mg: VT-1161 1200mg once daily for 4 days, then VT-1161 300mg once daily for 10 days
- Placebo: matching tablets over-encapsulated for blinding purposes
Period: Overall Study
Arm/Group | VT-1161 200/50mg | VT-1161 600/150mg | VT-1161 1200/300mg | Placebo
Started | 12 | 12 | 14 | 12
Completed | 9 | 11 | 11 | 12
Not Completed | 3 | 1 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VT-1161 200/50mg | VT-1161 600/150mg | VT-1161 1200/300mg | Matching Placebo | Total
Number analyzed (Participants) | 12 | 12 | 14 | 12 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (12.84) | 40.6 (11.71) | 34.05 (12.02) | 35.2 (10.27) | 38.9 (12.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 3 | 5 | 13
  Male | 9 | 10 | 11 | 7 | 37

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Therapeutic Cure at 42 Days for All-analysis Population
Description: For this trial, therapeutic cure was defined as clinical AND mycological cure. Clinical cure was defined as the absence of signs and symptoms of clinical disease. Mycological cure was defined as a negative KOH test and a negative fungal culture.
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | VT-1161 200/50mg | VT-1161 600/150mg | VT-1161 1200/300mg | Matching Placebo
Number analyzed (Participants) | 12 | 12 | 14 | 12
Participants | 2 | 1 | 3 | 0

ADVERSE EVENTS:
Arm/Group | VT-1161 200/50mg | VT-1161 600/150mg | VT-1161 1200/300mg | Matching Placebo
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/14 | 0/12
Other Adverse Events (participants affected / at risk) | 2/12 | 3/12 | 5/14 | 5/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VT-1161 200/50mg (N=12) | VT-1161 600/150mg (N=12) | VT-1161 1200/300mg (N=14) | Matching Placebo (N=12)
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Herpes Zoster (Infections and infestations) | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 1 | 0
Oral Herpes (Infections and infestations) | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1
Tooth Infection (Infections and infestations) | 0 | 0 | 1 | 0
Blood Pressure Increased (Investigations) | 0 | 1 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Ectopic Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1
Pyuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Paranasal Sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Neither institution nor principal investigator shall publish the results of the trial without prior written consent of the sponsor, which it may withhold in its sole discretion.